CLINICAL TRIAL: NCT02700373
Title: A Phase I, Single-Center, Double-Blind, Randomized, Single Ascending Dose Study of PDC-APB in Healthy Volunteers
Brief Title: A Phase I, Single-Center Study of PDC-APB in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hapten Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PDC-APB-CL01
Record Dates: First submitted 2016-02-19; First posted 2016-03-07 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Contact Dermatitis
MeSH Terms: conditions — Dermatitis, Contact | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PDC-APB (Experimental): PDC-APB Intra-Muscular (IM)
  One single dose will be administered with an inpatient direct observational period of 24 hours following the dose, followed by outpatient follow-up for a total of 28 days. After Day 28, the subject will continue to be followed up for study related AE assessments thru Week 24.
  Interventions: Drug: PDC-APB
- Placebo (Placebo Comparator): Placebo
  One single dose will be administered with an inpatient direct observational period of 24 hours following the dose, followed by outpatient follow-up for a total of 28 days. After Day 28, the subject will continue to be followed up for study related AE assessments thru Week 24.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PDC-APB
  Other Names: Active
  Arms: PDC-APB
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, single ascending dose study to assess the safety and tolerability of PDC-APB by intramuscular (IM) injection compared to placebo.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, single ascending dose study to assess the safety and tolerability of PDC-APB by intramuscular (IM) injection compared to placebo. In this First-in-Human study it is anticipated that up to 5 dose levels (2.5 mg, 10 mg, 0.125 mg, .375 mg and 1.0 mg PDC-APB) will be studied in sequential cohorts. Each cohort will enroll 8 subjects, 6 subjects randomized to active treatment and 2 randomized to placebo, in a double-blind manner. A sentinel group of 2 subjects in each cohort will be randomized to active (1 subject) or placebo (1 subject). If the dose is tolerated in the sentinel group, the remaining 6 subjects in the cohort will be treated (5 active and 1 placebo).

Safety will be assessed in each cohort before starting treatment at the next higher dose level. If the study treatment is tolerated and there are no findings that necessitate stopping the study, the next cohort will be treated at the next higher dose level, in the same manner. This process will continue until the highest intended dose (1 mL) is reached, or side effects that limit further dose escalation are observed.

ELIGIBILITY:
Inclusion Criteria:

Subjects are required to meet the following criteria in order to be included in the study:

1. Healthy male and female subjects as determined by medical history and physical examination, from 18 to 55 years of age, inclusive
2. History of previous exposure to poison ivy, oak, or sumac without development of significant contact dermatitis. Significant contact dermatitis is defined as a skin reaction that covered more than 10% of body surface area by the subject's estimation, occurred on the face or genitals, was rated by the subject as moderate or severe, or required treatment with topical, oral, or injectable (systemic) steroids for resolution of symptoms. History of exposure will be documented using the Allergic Contact Dermatitis Questionnaire (Appendix 1).
3. For female subjects: Surgically sterile or menopausal (at least 1 year absence of vaginal bleeding or spotting) and as confirmed by follicle-stimulating hormone (FSH) ≥ 40 mIU/mL. Females of childbearing age/potential may be included provided that they are using medically acceptable methods of birth control for 1 month prior to and for the duration of the study and for 3 months thereafter. Dual methods must be used, for example a hormonal method used with a barrier method.
4. For male subjects and their partners of childbearing potential: Willing to use two methods of contraception, one of which must be a barrier method, for the duration of the study and for 3 months after the last dose of study drug, and agreed not to donate sperm for 3 months after the last dose of study drug
5. A body mass index (BMI) between 18 and 32 kg/m2 inclusive
6. Able to participate and willing to give written informed consent and to comply with the study restrictions

Exclusion Criteria:

1. History of significant contact dermatitis secondary to exposure to poison ivy, poison oak, or poison sumac, as defined in Inclusion Criteria #2 (above)
2. Positive breath test for alcohol or urine test for drugs of abuse as per local standard at screening, or a history of alcohol or drug abuse within the past 24 months
3. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV), or HIV clinical laboratory test
4. Administration of, or need for, any prescription drug within 21 days, or over-the-counter drugs (except acetaminophen and ibuprofen ≤ 1 g/day or multivitamins, which are permitted)
5. Any screening laboratory evaluation outside the laboratory reference range that is judged by the investigator to be clinically significant (including hepatic and renal panels, complete blood count, chemistry panel, and urinalysis)
6. History of significant renal or urinary disease or active symptoms of renal or urinary disease. A history of renal stones or of urinary tract infections does not exclude a subject.
7. History of significant hepatic disease or impairment, or any active symptoms of hepatic disease
8. Presence of clinically significant gastrointestinal (GI) disorder or symptoms of active GI disease. A history of appendectomy of cholecystectomy does not exclude a subject.
9. History of significant cardiovascular disease, such as hypertension requiring drug therapy, congestive heart failure, stroke, angina, arrhythmias, or symptoms or signs of active cardiovascular disease, or a clinically significant abnormality on the screening ECG that the Sponsor considers unacceptable
10. History of significant psychiatric disease, including but not limited to: bipolar disorder, depression, anxiety, panic attacks, and schizophrenia
11. History or symptoms of significant central nervous system (CNS) disease, including but not limited to: transient ischemic attack (TIA), stroke, seizure disorder, history of loss of consciousness or head trauma, or behavioral disturbances
12. History of suicide attempt or report of suicidal ideation
13. Concomitant disease or any organ system condition or abnormality that could pose an unacceptable risk to the subject in this study, in the opinion of the investigator, based on possible interference with absorption, distribution, metabolism, or elimination of the study drug or possible effect of the study drug on the condition or abnormality
14. History of significant allergies requiring treatment with steroids (by topical or oral administration), or use in the previous year of any immunosuppressants or immunotherapy, or use of oral or topical antihistamines in the previous 14 days
15. Known or suspected allergy or cutaneous sensitivity to any product components, including sesame or sesame oil, benzyl alcohol, or ethanol
16. History of asthma, including subjects with asthma who require acute or maintenance inhaled or oral steroid use for control of symptoms, as well as subject with intermittent asthma who do not require corticosteroids.
17. History of any acute or chronic skin condition (except contact dermatitis as noted in Inclusion Criteria #2) or the presence of any rashes at screening or baseline.
18. Participation in an investigational drug or device study within 30 days prior to screening
19. Donation of blood over 400 mL within 60 days prior to screening and/or hemoglobin <7 mmol/L, or any plasma donation within 7 days prior to screening
20. Unwillingness or inability to comply with the study protocol for any reason

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Primary outcome measure for this study will be the overall safety profile observed during the post-treatment observation period in the study population. AEs will be classified by organ class using the coding system and by severity (Grade 1-4). | 24 Weeks
  The primary objective of the study is to assess the safety and tolerability of PDC-APB following single doses administered intramuscularly to healthy subjects between 18 and 55 years of age.

SECONDARY OUTCOMES:
Exposure to PDC-APB in study subjects. | 28 days
  The exploratory objective of the study is to document exposure of PDC-APB in study subjects by obtaining a small number of plasma samples following administration of PDC-APB by the IM route.

CONTACTS AND LOCATIONS:
Overall Officials: Chad S Boomershine, MD, Principal Investigator — Clinical Research Solutions
Locations (1):
- Clinical Research Solutions, Franklin, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes